CLINICAL TRIAL: NCT03932227
Title: EVAluation of the Non Inferiority of Interpretability of Cardiokin Compared to Holter
Acronym: EVANI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BioSerenity (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 2019-A00922-55
Record Dates: First submitted 2019-04-19; First posted 2019-04-30 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Electrocardiography, Ambulatory

STUDY DESIGN:
Intervention Model Description: Monocentric, cross study, randomized
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cardioskin-Holter (Other): Subjects in the randomized group A, start by wear the Cardioskin during 24h, and after wear the Holter during 24h.
  Interventions: Device: Cardioskin; Device: Holter
- Holter-Cardioskin (Other): Subjects in the randomized group B, start by wear the Holter during 24h, and after wear the Cardioskin during 24h.
  Interventions: Device: Cardioskin; Device: Holter

INTERVENTIONS:
Device: Cardioskin — Subjects will have a 24h recording with Cardioskin, next will be unequipped.
Device: Holter — Subjects will have a 24h recording with Holter, next will be unequipped.

SUMMARY:
The aim is to evaluate the electrocardiogram quality signal of the Cardioskin device and compare it with a Holter signal. For that, volunteers subjects will wear the Cardioskin and Holter, non-simultaneously, for about 24 hours.

This study is open, and will be carried out according to a cross plan. The trial will include approximately 36-40 subjects between 18 and 70 years old.

DETAILED DESCRIPTION:
The wear of the first device will be randomized. Each subject will wear the two devices.

One group will start with a 24-hour environmental recording with Cardioskin and then will perform another recording of about 24 hours with the Holter. Conversely, group B will start with the Holter and then will continue with Cardioskin. It is a randomization software that will assign a group to each included participant.

Each participant will come three times at hospital : one for inclusion and equipment of the first device, another to be unequipped and equipped of the second device. They will come another time to bring back the material. The total time of participation is of two days and half.

The first aim is to evaluate if the signal interpretability is non-inferior to an Holter, for a recording of 24h (classic analysis of rhythm).

The second aim is to evaluate if the 24 hours signal interpretability is non-inferior to an Holter in the case of a repolarization analysis.

The third aim is to compare the comfort and usability between Cardioskin and Holter.

ELIGIBILITY:
Inclusion Criteria:

* people between 18 and 70 years old

Exclusion Criteria:

* Minors
* Pregnant, parturient or breastfeeding women
* Refusal of consent
* Participant with known cardiac history
* Participant with cardiac arrhythmia observed during control ECG
* Participant who may be exposed to ionizing or electromagnetic radiation on days when devices (Cardioskin, Holter) will be worn
* Allergy to one of the components of the Cardioskin T-shirt, including:

Polyamide - Polyester - Elastane - Other synthetic materials - Silicone - Silver

* Allergy to one of the components of the electrodes used for the Holter (Kendall 530 or similar)
* Sensory disturbances that make the participant unresponsive to pain
* Motor or mental disorders that prevent the participant from expressing their pain -Behavioral problems that make the participant excessively Agitated or Aggressive
* Cardiorespiratory disorders that may be aggravated by mild compression of the chest
* Weight and / or size not suitable for the proposed Cardioskin T-shirt designs
* Open wound on the skin in the area covered by Cardioskin textile or by the electrodes of the Holter
* Irritation, and / or erythema in the area covered by the Cardioskin textile or by the electrodes of the Holter
* Pregnancy clinically detectable or known to a participant
* Participant with a high infectious risk
* Person wearing breast prostheses
* Simultaneous participation in another search

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2019-07-08 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
interpretability of signal | 48 hours
  The quality signal will be assess blindly by rythm specialists. For that,specialists will show is the isoelectric line is stable (answer "Yes" "No")
interpretability of signal | 48 hours
  The quality signal will be assess blindly by rythm specialists. For that,specialists will show the p waves are visible (answer "Yes" "No")
interpretability of signal | 48 hours
  The quality signal will be assess blindly by rythm specialists. For that,specialists will show if the R pic are visible (answer "Yes" "No")
interpretability of signal | 48 hours
  The quality signal will be assess blindly by rythm specialists. For that,specialists will show is the RR intervals are visible (answer "Yes" "No")
interpretability of signal | 48 hours
  Cardiac observations will lead to a unique evaluation of the quality signal: either "interpretable" either "non-interpretable" (answer "Yes" "No")

SECONDARY OUTCOMES:
interpretability of signal for a fine analysis of cardiac repolarization | 48 hours
  The quality signal will be assess blindly by rythm specialists. For that, specialists will observe if the QRS width is measurable (answer "Yes" "No")
interpretability of signal for a fine analysis of cardiac repolarization | 48 hours
  The quality signal will be assess blindly by rythm specialists. For that, specialists will observe if the T waves are visible (answer "Yes" "No")
interpretability of signal for a fine analysis of cardiac repolarization | 48 hours
  The quality signal will be assess blindly by rythm specialists. For that, specialists will observe if the ST segment is analyzable (answer "Yes" "No")
interpretability of signal for a fine analysis of cardiac repolarization | 48 hours
  The quality signal will be assess blindly by rythm specialists. For that, specialists will observe if the QT interval is measurable (answer "Yes" "No")
interpretability of signal for a fine analysis of cardiac repolarization | 48 hours
  These cardiac observations will lead to a unique evaluation of the quality signal: either "interpretable" either "non-interpretable" (answer "Yes" "No")
evaluation of comfort | 24 hours
  At the end of each recording, a subject will answer to a questionnary For comfort of the textile: Score of 0 to 70 points where 0 is comfortable and 70 is not comfortable.
evaluation of usability | 24 hours
  At the end of each recording, a subject will answer to a questionnary
  For usability of the system: score of 0 to 100 points where 0 is a bad usability and 100 is excellent

CONTACTS AND LOCATIONS:
Locations (1):
- European Hospital George Pompidou, Paris, France

IPD SHARING:
Plan to Share IPD: No